CLINICAL TRIAL: NCT00594503
Title: Hyperbaric Oxygen Therapy and SPECT Brain Imaging in Traumatic Brain Injury
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Paul G. Harch, M.D. (Other)
Collaborators: Harch Hyperbaric Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Paul G. Harch, M.D., Clinical Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Organization: Louisiana State University Health Sciences Center in New Orleans (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LSU IRB #6625
Record Dates: First submitted 2008-01-03; First posted 2008-01-15 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Residual Neurological, Cognitive, Emotional, Behavioral Effects From Traumatic Brain Injury
Keywords: traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hyperbaric oxygen therapy-TBI (Experimental): Low pressure hyperbaric oxygen therapy
  Interventions: Drug: Hyperbaric oxygen therapy

INTERVENTIONS:
Drug: Hyperbaric oxygen therapy — Total body exposure to increased atmospheric pressure oxygen

SUMMARY:
Hypothesis: That SPECT brain imaging tracks and is consistent with clinical improvements in patients receiving hyperbaric oxygen therapy (HBOT) for chronic traumatic brain injury.

DETAILED DESCRIPTION:
The study is a retrospective chart review of patients with chronic neurological, emotional, social, and cognitive deficits from mild, moderate, or severe traumatic brain injury who underwent SPECT brain imaging as part of their evaluation and treatment with hyperbaric oxygen therapy in my practice over the last two decades. The purpose of the study is to see if the functional imaging is consistent with the clinical and cognitive testing.

ELIGIBILITY:
Inclusion Criteria:

* Adults or children with traumatic brain injury at least one year old

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2007-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
SPECT brain imaging | After completion of HBOT
  Only for those subjects in which SPECT brain imaging was performed before hyperbaric oxygen therapy

SECONDARY OUTCOMES:
Clinical history and physical exam | After completion of HBOT
Cognitive testing | After the final HBOT
  Only for those subjects in which neuropsychological cognitive testing was performed before hyperbaric oxygen therapy

CONTACTS AND LOCATIONS:
Overall Officials: Paul G Harch, M.D., Principal Investigator — LSU School of Medicine, New Orleans
Locations (1):
- Family Physicians Center, Marrero, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No